CLINICAL TRIAL: NCT05427461
Title: Circulating " Cancer Cells / Macrophage " HYbrid Cells in Patients With Sarcoma, Part 2
Acronym: SAMHY2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Fondation ARC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22 SARC 03
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Leiomyosarcoma
Keywords: Leiomyosarcoma; Cancer cell/macrophage hybrid cells; Hybrid cells
MeSH Terms: conditions — Leiomyosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with leiomyosarcoma (Other)
  Interventions: Other: Blood samples will be collected at different times.

INTERVENTIONS:
Other: Blood samples will be collected at different times. — For patients with localized leiomyosarcoma, samples will be collected:
  * At Baseline.
  * Before surgery (for patients who have had neoadjuvant treatment (external radiotherapy and/or chemotherapy)).
  * After surgery.
  * At each control visit.
  * At local or metastatic recurrence (or at 24 months post inclusion if no progression).
  For patients with metastatic leiomyosarcoma, samples will be collected:
  * At Baseline.
  * At each therapeutic line.
  * At progression (or at 24 months post inclusion if no progression).

SUMMARY:
Pilot, prospective, monocentric study aimed at evaluating the rate of patients with circulating "cancer cell/macrophage" hybrid cells in the peripheral blood and the evolution of this rate over time.

The study will be conducted on a population of patients with leiomyosarcoma and treated in the context of routine care. 20 patients will be included:

* 10 patients with localized disease.
* 10 patients with metastatic disease.

For each included patient, blood samples will be collected during baseline visit and up to 24 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with leiomyosarcoma.
2. Diagnosis of sarcoma histologically confirmed by the RRePS network (Réseau de Référence en Pathologie des Sarcomes et des Viscères)
3. Localized or metastatic disease
4. Newly diagnosed patient who has not yet initiated specific treatment for sarcoma
5. Age ≥ 18 years
6. Patient affiliated to a Social Security system in France.
7. Patient having signed informed consent prior to inclusion in the study and prior to any specific study procedures

Exclusion Criteria:

1. Diagnosis of any other histological subtype of soft tissue sarcoma
2. Associated pathology(ies) that may interfere with the study procedure
3. Pregnant or breastfeeding woman
4. Any psychological, family, geographical or sociological condition that does not allow for compliance with the medical follow-up and/or procedures provided for in the study protocol.
5. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The longitudinal evolution of rate of patients with "cancer cell / macrophage" hybrid cells in peripheral blood. | 24 months after the end of inclusions.

SECONDARY OUTCOMES:
Quantification of circulating hybrid cells in peripheral blood by automatic measurement (Cell Counter Corning) and expressed in number of cells / millilitre of blood. | 24 months after the end of inclusions.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse, France